CLINICAL TRIAL: NCT02162810
Title: Effect of Steroids on Post-Operative Complications Following Proximal Hypospadias Repair
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We were unable to meet our enrollment goal necessary to analyze the outcome measures.
Sponsor: Francis Schneck (Other)
Responsible Party: Sponsor-Investigator, Francis Schneck, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: PRO14010275
Record Dates: First submitted 2014-03-11; First posted 2014-06-13 (Estimated); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Hypospadias
Keywords: hypospadias
MeSH Terms: conditions — Hypospadias | interventions — Prednisolone; Steroids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral steroids (Active Comparator): Systemic high-dose steroids (30 mg/kg methylprednisolone) have been shown in a randomized, double-blind, placebo-controlled trial in humans not to negatively impact wound infection or dehiscence rates, instead benefitting patients in the postoperative period in ways such as decreasing pain. An acute course of oral systemic steroids has been routinely used in patients under the age of 12 with asthma exacerbations (liquid prednisolone at 1-2 mg/kg/day in 1-2 divided doses for up to 10 days, although usually given for 5 days, which is at least 19 times less than the dose proven to be safe in the randomized controlled trial mentioned above) and proven to be safe without adverse effects. Effect of prednisolone on the systemic response and wound healing after colonic surgery.
  Interventions: Drug: Prednisolone
- placebo-controlled (Placebo Comparator): Simple Syrup will be used as the placebo
  Interventions: Drug: placebo-controlled

INTERVENTIONS:
Drug: Prednisolone — In order to analyze the data, we will establish a chart which will show the degree of cosmetic appearance, incidences and degree of complications. This we be assessed on a mild to severe scale.
  Other Names: Steroid
  Arms: oral steroids
Drug: placebo-controlled — In order to analyze the data, we will establish a chart which will show the degree of cosmetic appearance, incidences and degree of complications. This we be assessed on a mild to severe scale.
  Other Names: Unknowen
  Arms: placebo-controlled

SUMMARY:
The primary objective of this study is to determine the efficacy of administering a course of postoperative oral steroids in pediatric patients undergoing proximal hypospadias repair as prevention against complications. Specifically, the study aims to assess if the steroids i) decrease the incidence of wound breakdown, fistula formation, stenosis or stricture formation, and the need for subsequent redo-hypospadias surgeries and/or fistula repairs and ii) improve the quality of wound healing including the overall cosmetic appearance of the phallus (i.e. location of the urethral meatus).

DETAILED DESCRIPTION:
Hypospadias repair is a surgery that is, unfortunately, fraught with a high complication rate with problems that include urethrocutaneous fistula formation, complete wound breakdown, glans dehiscence, urethral diverticulum formation, retraction of the urethral meatus, urethral stricture, and meatal stenosis . Failure of a proximal hypospadias repair (i.e. the development of a post-operative complication) is unpredictable, and few modifiable risk factors having been identified. Complications necessitate subsequent surgical intervention for pediatric patients, which must be carried out under general anesthesia. Evidence regarding the harms of multiple general anesthetics for children is increasing. Additionally, with each surgical revision comes the morbidity associated with another post-surgical convalescence. Thus, any measure that can be gained as a way to increase the rate of success of proximal hypospadias repair would be of help to all pediatric urologists and patients with hypospadias. The proposed intervention of administering a 5 day course of placebo versus oral steroids at a dose equivalent to what is given for outpatient treatment of asthma exacerbations, is expected to have very low risk. This would be the only variation from the current practice and one that has never been studied in the past. Thus, it would be worthwhile to perform use scientific methods to determine if the administration of a short course of oral steroids is of benefit to healing and minimization of post-operative complications for hypospadias patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing proximal hypospadias repair

Exclusion Criteria:

* All patients currently taking steroids at the time of surgery or during the six-week recovery period as well as patients with betamethasone hypersensitivity will be excluded from the study. Selection will be based on parent willingness to allow the child to participate in the study.

Ages: 3 Months to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2014-05; Primary Completion 2022-05 (Actual); Study Completion 2022-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Schneck, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Steroids | Placebo-controlled
Started | 17 | 11
Completed | 12 | 10
Not Completed | 5 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — patients did not report compliance | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Steroids | Placebo-controlled | Total
Number analyzed (Participants) | 17 | 11 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 11 | 28
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 17 | 11 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 11 | 28
NICU Stay [Count of Participants; unit: Participants] | 11 | 5 | 16
Incidence of Comorbidities [Count of Participants; unit: Participants] | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Complication Rate After Hypospadias Repair
Description: Post-operative incidence of wound breakdown, fistula formation, stenosis or stricture formation, and the need for subsequent redo-hypospadias surgeries and/or fistula repairs, after Hypospadias repair.
Time Frame: postoperative follow up 7-12 days after the surgery following completion of the 5-day course of prednisolone vs. placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Steroids | Placebo-controlled
Number analyzed (Participants) | 17 | 11
Participants
  meatal retraction | 1 | 0
  meatal stenosis | 0 | 0
  glans dehiscence | 0 | 1
  skin breakdown along suture lines, urethra intact | 0 | 0
  urethra breakdown proximal to glans | 0 | 0
  urethrocutaneous fistula | 2 | 0
  suspected stricture | 0 | 0
  suspected urethral diverticulum | 1 | 0
Statistical Analysis 1: Comparison: Oral Steroids vs Placebo-controlled; Due to the number of 0 cell counts, it is not possible to do individual statistics for each complication, so we looked at the incidence of complications overall between the two arms; Test type: Other; p < .62, Fisher Exact

2. Primary Outcome: Meatus Location After Hypospadias Repair
Description: The overall cosmetic appearance of the phallus (i.e. location of the urethral meatus) post-operatively.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Steroids | Placebo-controlled
Number analyzed (Participants) | 17 | 11
Participants
  glanular | 13 | 8
  coronal | 0 | 0
  subcoronal | 0 | 0
  distal shaft | 0 | 0
  proximal shaft | 0 | 0
  penoscrotal | 4 | 2
  other | 0 | 1
Statistical Analysis 1: Comparison: Oral Steroids vs Placebo-controlled; Test type: Other; p < 0.61, Fisher Exact

3. Primary Outcome: Improvement of Chordee After Hypospadias Repair
Description: Improvement of Chordee post-operatively after Hypospadias repair.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Steroids | Placebo-controlled
Number analyzed (Participants) | 17 | 11
Participants
  improvement of chordee with degloving: resolved | 2 | 2
  improvement of chordee with degloving: improved | 3 | 1
  improvement of chordee with degloving: improvement described but not documented | 1 | 0
  improvement of chordee with degloving: no improvement | 8 | 7
  improvement of chordee with degloving: not described | 3 | 1
  improvement in ventral chordee: resolved | 2 | 0
  improvement in ventral chordee: improved | 2 | 2
  improvement in ventral chordee: improvement described but not documented | 0 | 0
  improvement in ventral chordee: no improvement | 5 | 2
  improvement in ventral chordee: not described | 8 | 7
  improvement of chordee with plication: resolved | 7 | 6
  improvement of chordee with plication: improved | 1 | 1
  improvement of chordee with plication: improvement described but not documented | 0 | 0
  improvement of chordee with plication: no improvement | 0 | 0
  improvement of chordee with plication: not described | 9 | 4
Statistical Analysis 1: Comparison: Oral Steroids vs Placebo-controlled; Improvement category: Chordee with Degloving; Test type: Other; p < .87, Fisher Exact
Statistical Analysis 2: Comparison: Oral Steroids vs Placebo-controlled; Improvement category: Ventral Chordee; Test type: Other; p < .64, Fisher Exact
Statistical Analysis 3: Comparison: Oral Steroids vs Placebo-controlled; Improvement category: Chordee with Plication; Test type: Other; p < .85, Fisher Exact

4. Primary Outcome: Complication Rate After Hypospadias Repair
Description: as for outcome 1
Time Frame: after stent removal at 4-12 weeks
Population: Further statistical analyses were not conducted on the data due to insufficient enrollment and follow-up participation, resulting in study termination.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Steroids | Placebo-controlled
Number analyzed (Participants) | 14 | 10
Participants
  meatal retraction | 1 | 0
  meatal stenosis | 0 | 0
  glans dehiscence | 0 | 1
  skin breakdown along suture lines, urethra intact | 0 | 0
  urethra breakdown proximal to glans | 0 | 0
  urethrocutaneous fistula | 2 | 0
  suspected stricture | 0 | 0
  suspected urethral diverticulum | 0 | 0

5. Primary Outcome: Meatus Location After Hypospadias Repair
Description: Post operative follow-up after stent removal at 4-12 weeks of the overall cosmetic appearance of the phallus (i.e. location of the urethral meatus).
Time Frame: after stent removal at 4-12 weeks
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Steroids | Placebo-controlled
Number analyzed (Participants) | 14 | 10
Participants
  glanular | 9 | 8
  coronal | 1 | 1
  subcoronal | 0 | 0
  distal shaft | 0 | 0
  proximal shaft | 0 | 0
  penoscrotal | 3 | 2
  other | 0 | 0

6. Secondary Outcome: Complications After Hypospadias Repair
Description: 6-month follow-up incidence of wound breakdown, fistula formation, stenosis or stricture formation, and the need for subsequent redo-hypospadias surgeries and/or fistula repairs, after Hypospadias repair.
Time Frame: 6 months after surgery
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Steroids | Placebo-controlled
Number analyzed (Participants) | 7 | 3
Participants
  meatal retraction | 0 | 0
  meatal stenosis | 0 | 0
  glans dehiscence | 0 | 0
  skin breakdown along suture lines, urethra intact | 0 | 0
  urethra breakdown proximal to glans | 0 | 0
  urethrocutaneous fistula | 2 | 1
  suspected stricture | 0 | 0
  suspected urethral diverticulum | 1 | 0

7. Secondary Outcome: Meatus Location After Hypospadias Repair
Description: The overall cosmetic appearance of the phallus (i.e. location of the urethral meatus) 6 months post-operatively.
Time Frame: 6-months after surgery
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Steroids | Placebo-controlled
Number analyzed (Participants) | 7 | 3
Participants
  glanular | 4 | 1
  coronal | 0 | 1
  subcoronal | 0 | 0
  distal shaft | 0 | 0
  proximal shaft | 0 | 0
  penoscrotal | 3 | 1
  other | 0 | 0

8. Secondary Outcome: Healing Outcomes After Hypospadias Repair, Follow up After Toilet Training
Description: i) the incidence of wound breakdown, fistula formation, stenosis or stricture formation, and the need for subsequent redo-hypospadias surgeries and/or fistula repairs and ii) the quality of wound healing including improvement of Chordee, and the overall cosmetic appearance of the phallus (i.e. location of the urethral meatus). Late complications can occur. Therefore, this needs to be evaluated at the specified interval. This is the standard of care at Children's Hospital of Pittsburgh of UPMC Pediatric Urology department.
Time Frame: Approximately at 4 years of age
Population: The study was terminated prior to the 4 year follow up due to lack of sufficient patient data to analyze; therefore, there was no post-toilet training follow up data collected.
Arm/Group | Oral Steroids | Placebo-controlled
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months post-op.
Arm/Group | Oral Steroids | Placebo-controlled
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/11
Other Adverse Events (participants affected / at risk) | 0/17 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/10/NCT02162810/Prot_SAP_000.pdf